CLINICAL TRIAL: NCT02577289
Title: Evaluation of Bone Quantity in Open Sinus Lift Technique With Simultaneous Implantation Using Platelet Rich Fibrin (PRF) Versus Nano-crystalline Hydroxyapatite as Sole Grafting Material in Patients With Atrophied Posterior Maxillary Ridge
Brief Title: Open Sinus Lift Technique With Simultaneous Implantation Using Platelet Rich Fibrin (PRF) Versus Nano-crystalline Hydroxyapatite
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, waleed Mohamed Mohamed Mahmoud nour el din, Master student, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: open_sinus_augmentation
Record Dates: First submitted 2015-10-13; First posted 2015-10-16 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Atrophied Posterior Maxillary Ridge
Keywords: simultaneous implantation; Dental implant; Open sinus Lifting; PRF; platelet rich fibrin (PRF)
MeSH Terms: interventions — Prolactin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group ( Hydroxyappetite) (Active Comparator): Patients will undergo open sinus lift using nano crystalline hydroxyapatite as augmentation material and placing implants simultaneously then evaluation of bone quantity in open sinus lift technique with simultaneous implantation ( Nano crystalline hydroxyapatite)
  Interventions: Procedure: Evaluation of bone quantity in open sinus lift technique with simultaneous implantation ( Nano crystalline hydroxyapatite)
- Test group (PRF) (Experimental): Patients will undergo open sinus lift using PRF as sole augmentation material and placing implants simultaneously then Evaluation of bone quantity in open sinus lift technique with simultaneous implantation (PRF)
  Interventions: Procedure: Evaluation of bone quantity in open sinus lift technique with simultaneous implantation (PRF)

INTERVENTIONS:
Procedure: Evaluation of bone quantity in open sinus lift technique with simultaneous implantation ( Nano crystalline hydroxyapatite) — • The sinus cavity will be augmented with bone graft ( Nano crystalline hydroxyapatite)
  Arms: Control group ( Hydroxyappetite)
Procedure: Evaluation of bone quantity in open sinus lift technique with simultaneous implantation (PRF) — platelet rich fibrin (PRF) as sole grafting material in created space (PRF)
  Arms: Test group (PRF)

SUMMARY:
Evaluation of bone quantity in open sinus lift technique with space maintaining using platelet rich fibrin (PRF) as sole augmentation material versus nano crystalline hydroxyapatite with simultaneous placing of implants.

DETAILED DESCRIPTION:
Evaluation of bone quantity in open sinus lift technique with simultaneous implantation using platelet rich fibrin (PRF) versus Nano-crystalline Hydroxyapatite as sole grafting material in patients with atrophied posterior maxillary ridge which provides a new modality for treatment of patients with atrophied posterior maxillary ridge with least cost and a much easier way using platelet rich fibrin (PRF) as substitution to bone graft

ELIGIBILITY:
Inclusion Criteria:

* All patients should be seeking for implant supported prosthesis in posterior maxilla bilaterally
* All patients should have atrophied posterior maxillary ridge with the maximum height of the alveolar bone is from 3 mm to 5 mm

Exclusion Criteria:

* Ongoing steroid therapy;
* Uncontrolled diabetes;
* Recent cardiovascular diseases;
* Inflammation of the maxillary sinus;
* Previous radiant therapy for neoplastic pathologies
* Patient who have had previous failed sinus augmentation, or exhibited pathological finding or had a history of maxillary sinus disease or operations or whose medical condition might increase surgical risk of the research protocol were excluded.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The amount of new bone formation the sinus cavity using CBCT | 6 months
  the amount of new bone formation of PRF in comparison with Nano-crystalline hydroxyappetite in millimeters using cone beam computed tomography (CBCT)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of oral and dental medicine, Cairo, Cairo Governorate, Egypt

REFERENCES:
- [Background] Jemt T, Lekholm U. Implant treatment in edentulous maxillae: a 5-year follow-up report on patients with different degrees of jaw resorption. Int J Oral Maxillofac Implants. 1995 May-Jun;10(3):303-11. PMID 7615326
- [Background] Raghoebar GM, Batenburg RH, Timmenga NM, Vissink A, Reintsema H. Morbidity and complications of bone grafting of the floor of the maxillary sinus for the placement of endosseous implants. Mund Kiefer Gesichtschir. 1999 May;3 Suppl 1:S65-9. doi: 10.1007/PL00014520. PMID 10414086
- [Background] Misch CE. Implant design considerations for the posterior regions of the mouth. Implant Dent. 1999;8(4):376-86. doi: 10.1097/00008505-199904000-00008. PMID 10709483
- [Background] Lundgren S, Andersson S, Gualini F, Sennerby L. Bone reformation with sinus membrane elevation: a new surgical technique for maxillary sinus floor augmentation. Clin Implant Dent Relat Res. 2004;6(3):165-73. PMID 15726851
- [Background] Sohn DS, Lee JS, Ahn MR, Shin HI. New bone formation in the maxillary sinus without bone grafts. Implant Dent. 2008 Sep;17(3):321-31. doi: 10.1097/ID.0b013e318182f01b. PMID 18784532
- [Background] Dohan DM, Choukroun J, Diss A, Dohan SL, Dohan AJ, Mouhyi J, Gogly B. Platelet-rich fibrin (PRF): a second-generation platelet concentrate. Part III: leucocyte activation: a new feature for platelet concentrates? Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Mar;101(3):e51-5. doi: 10.1016/j.tripleo.2005.07.010. PMID 16504851
- [Background] Sakka S, Coulthard P. Bone quality: a reality for the process of osseointegration. Implant Dent. 2009 Dec;18(6):480-5. doi: 10.1097/ID.0b013e3181bb840d. PMID 20009601
- [Background] Dohan DM, Choukroun J, Diss A, Dohan SL, Dohan AJ, Mouhyi J, Gogly B. Platelet-rich fibrin (PRF): a second-generation platelet concentrate. Part I: technological concepts and evolution. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Mar;101(3):e37-44. doi: 10.1016/j.tripleo.2005.07.008. Epub 2006 Jan 19. PMID 16504849
- [Background] Dohan DM, Choukroun J, Diss A, Dohan SL, Dohan AJ, Mouhyi J, Gogly B. Platelet-rich fibrin (PRF): a second-generation platelet concentrate. Part II: platelet-related biologic features. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Mar;101(3):e45-50. doi: 10.1016/j.tripleo.2005.07.009. Epub 2006 Jan 10. PMID 16504850
- [Background] Choukroun J, Diss A, Simonpieri A, Girard MO, Schoeffler C, Dohan SL, Dohan AJ, Mouhyi J, Dohan DM. Platelet-rich fibrin (PRF): a second-generation platelet concentrate. Part IV: clinical effects on tissue healing. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Mar;101(3):e56-60. doi: 10.1016/j.tripleo.2005.07.011. PMID 16504852
- [Background] Cho JS, Ko YN, Koo HY, Kang YC. Synthesis of nano-sized biphasic calcium phosphate ceramics with spherical shape by flame spray pyrolysis. J Mater Sci Mater Med. 2010 Apr;21(4):1143-9. doi: 10.1007/s10856-009-3980-1. Epub 2010 Jan 6. PMID 20052521
- [Background] Ferraz MP, Monteiro FJ, Manuel CM. Hydroxyapatite nanoparticles: A review of preparation methodologies. J Appl Biomater Biomech. 2004 May-Aug;2(2):74-80. PMID 20803440
- [Background] 20. Best SM, Porter AE, Thian ES, Huang J: Bioceramics: Past, present and for the future. J Eur Ceram Soc 28: 1319, 2008.
- [Background] Bohner M, Baumgart F. Theoretical model to determine the effects of geometrical factors on the resorption of calcium phosphate bone substitutes. Biomaterials. 2004 Aug;25(17):3569-82. doi: 10.1016/j.biomaterials.2003.10.032. PMID 15020131
- [Background] von Doernberg MC, von Rechenberg B, Bohner M, Grunenfelder S, van Lenthe GH, Muller R, Gasser B, Mathys R, Baroud G, Auer J. In vivo behavior of calcium phosphate scaffolds with four different pore sizes. Biomaterials. 2006 Oct;27(30):5186-98. doi: 10.1016/j.biomaterials.2006.05.051. Epub 2006 Jun 21. PMID 16790273
- [Background] 23. Kalita SJ, Bhardwaj a, Bhatt H a: Nanocrystalline calcium phosphate ceramics in biomedical engineering. Mater Sci Eng CBiomimetic Supramol Sist 27: 441, 2007.
- [Background] Mazor Z, Mamidwar S. Effect of Nanocrystalline Calcium Sulfate Bone Graft in a Bilateral Sinus-Augmentation Procedure: A Case Report. Clin Adv Periodontics. 2015 Feb;5(1):76-81. doi: 10.1902/cap.2013.130022. PMID 32689744
- [Background] Mazor Z, Horowitz RA, Del Corso M, Prasad HS, Rohrer MD, Dohan Ehrenfest DM. Sinus floor augmentation with simultaneous implant placement using Choukroun's platelet-rich fibrin as the sole grafting material: a radiologic and histologic study at 6 months. J Periodontol. 2009 Dec;80(12):2056-64. doi: 10.1902/jop.2009.090252. PMID 19961389
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Result] Boyne PJ, James RA. Grafting of the maxillary sinus floor with autogenous marrow and bone. J Oral Surg. 1980 Aug;38(8):613-6. No abstract available. PMID 6993637
- [Result] Aghaloo TL, Moy PK. Which hard tissue augmentation techniques are the most successful in furnishing bony support for implant placement? Int J Oral Maxillofac Implants. 2007;22 Suppl:49-70. PMID 18437791
- [Result] Fugazzotto PA, Vlassis J. Long-term success of sinus augmentation using various surgical approaches and grafting materials. Int J Oral Maxillofac Implants. 1998 Jan-Feb;13(1):52-8. PMID 9509780
- [Result] Hurzeler MB, Kirsch A, Ackermann KL, Quinones CR. Reconstruction of the severely resorbed maxilla with dental implants in the augmented maxillary sinus: a 5-year clinical investigation. Int J Oral Maxillofac Implants. 1996 Jul-Aug;11(4):466-75. PMID 8803342
- [Result] Smiler DG, Johnson PW, Lozada JL, Misch C, Rosenlicht JL, Tatum OH Jr, Wagner JR. Sinus lift grafts and endosseous implants. Treatment of the atrophic posterior maxilla. Dent Clin North Am. 1992 Jan;36(1):151-86; discussion 187-8. PMID 1737600
- [Result] Chanavaz M. Maxillary sinus: anatomy, physiology, surgery, and bone grafting related to implantology--eleven years of surgical experience (1979-1990). J Oral Implantol. 1990;16(3):199-209. PMID 2098563
- [Result] Jaffin RA, Berman CL. The excessive loss of Branemark fixtures in type IV bone: a 5-year analysis. J Periodontol. 1991 Jan;62(1):2-4. doi: 10.1902/jop.1991.62.1.2. PMID 2002427